CLINICAL TRIAL: NCT03442608
Title: A Multi-center, Randomized, Controlled Trial to Investigate the Efficacy and Safety of Long-term Therapeutic Hypothermia in Adult Patients With Poor-grade Aneurysmal Subarachnoid Hemorrhage
Brief Title: Trial of Long-term Therapeutic Hypothermia for Poor-grade Aneurysmal Subarachnoid Hemorrhage
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Collaborators: First Affiliated Hospital of Fujian Medical University (Other); Central South University (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); Tang-Du Hospital (Other); First Affiliated Hospital of Harbin Medical University (Other); The First Hospital of Jilin University (Other); The First Affiliated Hospital of Dalian Medical University (Other); Shanxi Cardiovascular Hospital (Other); Qilu Hospital of Shandong University (Other); First Affiliated Hospital of Wenzhou Medical University (Other); Shandong Provincial Hospital (Other Government); Yantai Yuhuangding Hospital (Other); Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Ning Wang, Professor, Xuanwu Hospital, Beijing
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LTHSAH-1
Record Dates: First submitted 2018-01-16; First posted 2018-02-22 (Actual); Last update posted 2018-02-26 (Actual); Status verified 2018-02

CONDITIONS: Hypothermia; Aneurysmal Subarachnoid Hemorrhage
MeSH Terms: conditions — Hypothermia; Subarachnoid Hemorrhage

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mild hypothermia (Experimental): Device: Zoll 2000 and/or CureWrap 3500 cooling system,lasting 5 to 7 days, the core temperature will be controlled in 33-35 degree.
  Interventions: Procedure: Zoll 2000 and/or CureWrap 3500 cooling system
- northermia (Placebo Comparator): normal physical cooling methods,like ice bag, conditionally required.
  Interventions: Procedure: Zoll 2000 and/or CureWrap 3500 cooling system

INTERVENTIONS:
Procedure: Zoll 2000 and/or CureWrap 3500 cooling system — Device(Zoll 2000 and/or CureWrap 3500 cooling system),lasting 5 to 7 days, the core temperature will be controlled in 33-35 degree.

SUMMARY:
This study is a prospective, multi-centre, randomized,controlled trial to compare the efficacy of long-term mild hypothermia with normothermic intensive management in patients with poor-grade aneurysmal subarachnoid hemorrhage.

The primary hypothesis is that the induction of mild hypothermia (maintained at 32-35℃) for at least 5 days would improve the outcome of patients at six months post hemorrhage compared with normothermia.

DETAILED DESCRIPTION:
Aneurysmal subarachnoid hemorrhage (aSAH), especially poor-grade aSAH, is a medical emergency with very high morbidity and mortality rates. SAH constitutes a major public health concern in developed and developing countries. There were several clinical trials of hypothermia for aSAH conducted, however, with conflicting results.

Hypothermia therapy treatment is currently used in our department and other large neurosurgical centers across China to decrease the intracranial pressure (ICP), mitigate some of the destructive processes, and improve the functional outcome of patients with poor-grade aSAH. When the decision was made, the patients would be placed in wrapped cooling blankets or intravascular cooling device after they were sedated, intubated and mechanically ventilated. The patients would receive continuous infusions of some drugs using an infusion pump to prevent shivering. Once the patient's rectal, nasopharyngeal or blood temperature reached 32˚C, it was kept at approximately that temperature (32-35˚C) 3 to 7 days. Then the patients were passively rewarmed to a temperature of 36 to 37˚C at a rate no greater than 0.25˚C/hour, by gradual adjustment of the blanket thermostat.

The present multi-center, randomized controlled trials is designed to investigate the efficacy and safety of long-term (3 days) mild hypothermia versus normothermia on the outcome of patients with poor-grade aSAH. The primary outcome is the neurological function assessed at 1,3, 6 months post injury with the Glasgow Outcome Score (GOS). Additionally, the following data will also be recorded and compared: the baseline data, Glasgow Coma Score,imaging examination (e.g. CT scan), intracranial pressure, laboratory tests (e.g. blood routine test, liver and kidney function, blood gas analysis, etc), the complications (e.g. pneumonia, significant bleeding) and so on.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 65 years within 72 hours after subarachnoid hemorrhage;
* Neurosurgical clipping or coiling for aneurysm;
* Hunt-Hess IV-V scale;
* The intracranial pressure is more than 20 mmHg.

Exclusion Criteria:

* GCS of 3 with bilateral fixed and dilated pupils;
* No spontaneous breathing or cardiac arrest at the scene of hemorrhage;
* No consent;
* Pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-03-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Neurological function | 6 months after hemorrhage
  The neurological function will be evaluated at 6 months after hemorrhage by 2 specialized investigators who are unaware of the patients' allocation according to five-category Glasgow Outcome Scale as follows: 1, death; 2, vegetative state - unable to interact with the environment; 3, severe disability - unable to live independently but able to follow commands; 4, moderate disability - capable of living independently but unable to return to work or school; and 5, good recovery - able to return to work or school.

SECONDARY OUTCOMES:
Intracranial pressure | Admission, day 1, day 2, day 3, day 4, day 5, day 6, day 7, day 14, until the monitor is removed
  The effect of long-term hypothermia on ICP control will be determined.
Length of ICU stay | 6 months post hemorrhage
  The numbers of days in the ICU
Length of hospital stay | 6 months post hemorrhage
  The numbers of days in the hospital.
Frequency of complications | 6 months post hemorrhage
  Frequency of complications during the the study such as pneumonia, coagulation disturbance,electrolyte disturbances, liver and kidney function abnormality will be recorded and compared between groups.
Mortality rate | 6 months after hemorrhage
  The proportion of death will be determined

CONTACTS AND LOCATIONS:
Overall Officials: Ning Wang, MD,PhD, Principal Investigator — Xuanwu Hospital,Capital Medical University, Beijing

REFERENCES:
- [Background] Seule MA, Muroi C, Mink S, Yonekawa Y, Keller E. Therapeutic hypothermia in patients with aneurysmal subarachnoid hemorrhage, refractory intracranial hypertension, or cerebral vasospasm. Neurosurgery. 2009 Jan;64(1):86-92; discussion 92-3. doi: 10.1227/01.NEU.0000336312.32773.A0. PMID 19050656
- [Derived] Qu X, Shang F, Zhao H, Qi M, Cheng W, Xu Y, Jiang L, Chen W, Wang N, Zhang H. Targeted temperature management at 33 degrees Celsius in patients with high-grade aneurysmal subarachnoid hemorrhage: a protocol for a multicenter randomized controlled study. Ann Transl Med. 2021 Apr;9(7):581. doi: 10.21037/atm-20-4719. PMID 33987279